CLINICAL TRIAL: NCT02990338
Title: A Phase 3 Randomized, Open-label, Multicenter Study Comparing Isatuximab (SAR650984) in Combination With Pomalidomide and Low-Dose Dexamethasone Versus Pomalidomide and Low-Dose Dexamethasone in Patients With Refractory or Relapsed and Refractory Multiple Myeloma
Brief Title: Multinational Clinical Study Comparing Isatuximab, Pomalidomide, and Dexamethasone to Pomalidomide and Dexamethasone in Refractory or Relapsed and Refractory Multiple Myeloma Patients
Acronym: ICARIA-MM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC14335; U1111-1180-6262 (Registry Identifier: ICTRP); 2016-003097-41 (EudraCT Number)
Record Dates: First submitted 2016-12-04; First posted 2016-12-13 (Estimated); Results first posted 2019-12-06 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Plasma Cell Myeloma
Keywords: Anti-CD38 monoclonal antibody
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Pd (pomalidomide + dexamethasone) (Active Comparator): Participants received pomalidomide 4 milligrams (mg) Per os (PO) on Days 1 to 21 of each 28-day treatment cycle plus dexamethasone 40 mg (participants greater than or equal to (>=) 75 years of age received 20 mg dexamethasone) PO on Days 1, 8, 15 and 22 of each 28-day treatment cycle until disease progression or unacceptable toxicity or participant's wish to discontinue study treatment, or any other reason, whichever comes first (maximum exposure: 306.6 weeks).
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone
- IPd (isatuximab + pomalidomide + dexamethasone) (Experimental): Participants received isatuximab 10 milligrams per kilogram (mg/kg) intravenous (IV) infusion on Days 1, 8, 15, and 22 at Cycle 1, and then on Days 1 and 15 of subsequent cycles plus pomalidomide 4 mg PO on Days 1 to 21 of each 28-day treatment cycle and dexamethasone 40 mg (participants >= 75 years of age received 20 mg dexamethasone), PO or IV on Day 1, 8, 15, 22 of each 28-day treatment cycle until disease progression or unacceptable toxicity or participant's wish to discontinue study treatment, or any other reason, whichever comes first (maximum exposure: 311.0 weeks).
  Interventions: Drug: Isatuximab; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Isatuximab — Pharmaceutical form: solution for infusion Route of administration: intravenous
  Other Names: SAR650984; Sarclisa
  Arms: IPd (isatuximab + pomalidomide + dexamethasone)
Drug: Pomalidomide — Pharmaceutical form: capsule Route of administration: oral
  Other Names: POMALYST IMNOVID
Drug: Dexamethasone — Pharmaceutical form: tablets or solution for infusion Route of administration: oral or intravenous

SUMMARY:
Primary Objective:

To demonstrate the benefit of isatuximab in combination with pomalidomide and low-dose dexamethasone in the prolongation of Progression Free Survival (PFS) as compared to pomalidomide and low-dose dexamethasone in participants with refractory or relapsed and refractory multiple myeloma (MM).

Secondary Objectives:

* To evaluate the Overall Response Rate (ORR) as per International Myeloma Working Group (IMWG) criteria in each arm.
* To compare the Overall Survival (OS) between the two arms.
* To evaluate the Time To Progression (TTP) in each arm.
* To evaluate the PFS in high risk cytogenetic population in each arm.
* To evaluate the Duration of Response (DOR) in each arm.
* To evaluate the safety in both treatment arms.
* To determine the Pharmacokinetic profile of isatuximab in combination with pomalidomide.
* To evaluate the immunogenicity of isatuximab.
* To assess disease-specific and generic health-related quality of life (HRQL), disease and treatment-related symptoms, health state utility, and health status.

DETAILED DESCRIPTION:
The duration of the study for the participants included a period for screening of up to 21 days (or up to 28 days for women who can become pregnant). Participants continued study treatment until disease progression, unacceptable adverse reaction, participants' wish or other reason of discontinuation.

During follow-up, participants who discontinued the study treatment due to progression of the disease were followed every 3 months (12 weeks) for survival (or until cut-off date), and participants who discontinued the study treatment prior to documentation of disease progression were followed-up every 4 weeks until disease progression, and then every 3 months (12 weeks) for survival (or until cut-off date).

ELIGIBILITY:
Inclusion criteria :

* Age superior or equal to 18 years or country's legal age of majority if the legal age was superior to 18 years old.
* Participants had a documented diagnosis of multiple myeloma with evidence of measurable disease i.e. serum M protein superior or equal to 0.5 grams per decilitre (g/dL) measured using serum protein immunoelectrophoresis and or urine M protein superior or equal to 200 mg per 24 hours measured using urine protein immunoelectrophoresis.
* Participants had received at least 2 prior lines of anti-myeloma therapy, which must include at least 2 consecutive cycles of lenalidomide and a proteasome inhibitor (bortezomib, carfilzomib or ixazomib) given alone or in combination.
* Participants had failed treatment with lenalidomide and a proteasome inhibitor (bortezomib, carfilzomib, or ixazomib) alone or in combination (Intolerant, progression within 6 months after reaching Partial Response or better).
* Participants had progressed on or within 60 days after end of previous therapy before to study entry, i.e., refractory to the last line of treatment.

Exclusion criteria:

* Primary refractory multiple myeloma defined as participants who had never achieved at least a minimal response (MR) with any treatment during the disease course.
* Free Light Chain measurable disease only.
* Prior therapy with pomalidomide.
* Any anti-myeloma drug treatment within 14 days before randomization, including dexamethasone.
* Eastern Cooperative Oncology Group performance status superior to 2.
* Platelets inferior to 75 000 cells per microliter (mcL) if inferior to 50% of bone marrow (BM) nucleated cells are plasma cells, and inferior to 30 000 cells per mcL if superior or equal to 50% of BM nucleated cells are plasma cells. Platelet transfusion was not allowed within three days before the screening visit.
* Absolute neutrophil count inferior to 1000 per mcL (1*10^9/L).
* Creatinine clearance inferior to 30 mL per minute (Modification of Diet in Renal Disease [MDRD] Formula).
* Total bilirubin superior to 2*ULN (Upper Limit of Normal).
* Corrected serum calcium superior to 14 milligrams per deciliter (mg/dL) (superior to 3.5 millimoles per liter (mmol/L).
* Aspartate aminotransferase (AST) and/or Alanine Aminotransferase (ALT) superior to 3*ULN.
* Hypersensitivity to immunomodulatory drugs (IMiDs) (thalidomide or lenalidomide) defined as any hypersensitivity reaction leading to stop IMiDs within the 2 first cycles or toxicity, which does meet intolerance definition.
* Hypersensitivity to dexamethasone, sucrose histidine (as base and hydrochloride salt), and polysorbate 80 or any of the components of study therapy that are not amenable to premedication with steroids, or H2 blockers that would prohibit further treatment with these agents.
* Significant cardiac dysfunction; myocardial infarction within 12 months; unstable, poorly controlled angina pectoris.
* Pregnant or breastfeeding woman or female who intends to become pregnant during the participation in the study.
* Male participants who disagreed to practice true abstinence or disagreed to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and at least 3 or 5 months following study treatment discontinuation, even if he had undergone a successful vasectomy.
* All participants who disagreed to refrain from donating blood while on study treatment and for 4 weeks after discontinuation from this study treatment.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2018-11-22 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (111):
- United States (2):
  - BRCR Medical Center Inc. Site Number : 8400002, Plantation, Florida
  - Dana Farber Site Number : 8400006, Boston, Massachusetts
- Australia (5):
  - Investigational Site Number : 0360004, St Leonards, New South Wales
  - Investigational Site Number : 0360001, Waratah, New South Wales
  - Investigational Site Number : 0360005, Melbourne, Victoria
  - Investigational Site Number : 0360002, Melbourne, Victoria
  - Investigational Site Number : 0360006, Richmond, Victoria
- Belgium (4):
  - Investigational Site Number : 0560003, Antwerp
  - Investigational Site Number : 0560002, Brussels
  - Investigational Site Number : 0560004, Ghent
  - Investigational Site Number : 0560001, Leuven
- Canada (3):
  - Investigational Site Number : 1240001, Montreal, Quebec
  - Investigational Site Number : 1240004, Montreal, Quebec
  - Investigational Site Number : 1240005, Sherbrooke, Quebec
- Czechia (5):
  - Investigational Site Number : 2030005, Brno
  - Investigational Site Number : 2030004, Hradec Králové
  - Investigational Site Number : 2030001, Olomouc
  - Investigational Site Number : 2030002, Ostrava - Poruba
  - Investigational Site Number : 2030003, Prague
- Investigational Site Number : 2080002, Aalborg, Denmark
- France (19):
  - Investigational Site Number : 2500021, Bayonne
  - Investigational Site Number : 2500008, Caen
  - Investigational Site Number : 2500009, Dijon
  - Investigational Site Number : 2500017, Grenoble
  - Investigational Site Number : 2500013, La Roche-sur-Yon
  - Investigational Site Number : 2500003, Lille
  - Investigational Site Number : 2500023, Limoges
  - Investigational Site Number : 2500019, Montpellier
  - Investigational Site Number : 2500002, Nantes
  - Investigational Site Number : 2500015, Paris
  - Investigational Site Number : 2500016, Paris
  - Investigational Site Number : 2500005, Pessac
  - Investigational Site Number : 2500004, Pierre-Bénite
  - Investigational Site Number : 2500007, Poitiers
  - Investigational Site Number : 2500025, Reims
  - Investigational Site Number : 2500014, Rennes
  - Investigational Site Number : 2500001, Toulouse
  - Investigational Site Number : 2500012, Tours
  - Investigational Site Number : 2500018, Vandœuvre-lès-Nancy
- Investigational Site Number : 2760001, Leipzig, Germany
- Greece (5):
  - Investigational Site Number : 3000002, Athens
  - Investigational Site Number : 3000005, Athens
  - Investigational Site Number : 3000001, Athens
  - Investigational Site Number : 3000004, Pátrai
  - Investigational Site Number : 3000003, Thessaloniki
- Hungary (3):
  - Investigational Site Number : 3480001, Budapest
  - Investigational Site Number : 3480003, Budapest
  - Investigational Site Number : 3480002, Debrecen
- Italy (9):
  - Investigational Site Number : 3800001, Bologna
  - Investigational Site Number : 3800010, Catania
  - Investigational Site Number : 3800009, Florence
  - Investigational Site Number : 3800008, Genova
  - Investigational Site Number : 3800007, Milan
  - Investigational Site Number : 3800002, Milan
  - Investigational Site Number : 3800006, Padua
  - Investigational Site Number : 3800004, Terni
  - Investigational Site Number : 3800003, Torino
- Japan (8):
  - Investigational Site Number : 3920001, Nagoya, Aichi-ken
  - Investigational Site Number : 3920005, Shibukawa-shi, Gunma
  - Investigational Site Number : 3920004, Sapporo, Hokkaido
  - Investigational Site Number : 3920006, Kyoto, Kyoto
  - Investigational Site Number : 3920008, Suwa-shi, Nagano
  - Investigational Site Number : 3920003, Okayama, Okayama-ken
  - Investigational Site Number : 3920007, Sunto-gun, Shizuoka
  - Investigational Site Number : 3920002, Shibuya-ku, Tokyo
- New Zealand (4):
  - Investigational Site Number : 5540001, Takapuna, Auckland
  - Investigational Site Number : 5540004, Dunedin, Otago
  - Investigational Site Number : 5540003, Hamilton, Waikato Region
  - Investigational Site Number : 5540002, Auckland
- Investigational Site Number : 5780001, Oslo, Norway
- Poland (4):
  - Investigational Site Number : 6160005, Krakow, Lesser Poland Voivodeship
  - Investigational Site Number : 6160003, Lublin, Lubusz Voivodeship
  - Investigational Site Number : 6160001, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160002, Chorzów, Silesian Voivodeship
- Portugal (3):
  - Investigational Site Number : 6200004, Coimbra
  - Investigational Site Number : 6200002, Lisbon
  - Investigational Site Number : 6200001, Porto
- Russia (3):
  - Investigational Site Number : 6430004, Moscow
  - Investigational Site Number : 6430001, Moscow
  - Investigational Site Number : 6430002, Moscow
- Investigational Site Number : 7030001, Bratislava, Slovakia
- South Korea (5):
  - Investigational Site Number : 4100007, Hwasun-gun, Jeollanam-do
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100006, Incheon
  - Investigational Site Number : 4100005, Seoul
- Spain (6):
  - Investigational Site Number : 7240005, Santiago de Compostela, A Coruña [La Coruña]
  - Investigational Site Number : 7240001, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240006, Santander, Cantabria
  - Investigational Site Number : 7240002, Pamplona, Navarre
  - Investigational Site Number : 7240003, Madrid
  - Investigational Site Number : 7240004, Salamanca
- Sweden (2):
  - Investigational Site Number : 7520004, Luleå
  - Investigational Site Number : 7520005, Uddevalla
- Taiwan (4):
  - Investigational Site Number : 1580004, Kaohsiung City
  - Investigational Site Number : 1580002, Taichung
  - Investigational Site Number : 1580001, Taipei
  - Investigational Site Number : 1580003, Taoyuan District
- Turkey (Türkiye) (10):
  - Investigational Site Number : 7920001, Ankara
  - Investigational Site Number : 7920002, Antalya
  - Investigational Site Number : 7920005, Istanbul
  - Investigational Site Number : 7920006, Istanbul
  - Investigational Site Number : 7920003, Istanbul
  - Investigational Site Number : 7920004, Istanbul
  - Investigational Site Number : 7920008, Izmir
  - Investigational Site Number : 7920010, Izmir
  - Investigational Site Number : 7920009, Kayseri
  - Investigational Site Number : 7920007, Kocaeli
- United Kingdom (3):
  - Investigational Site Number : 8260002, London, London, City of
  - Investigational Site Number : 8260003, London, London, City of
  - Investigational Site Number : 8260001, London, London, City of

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Background] Attal M, Richardson PG, Rajkumar SV, San-Miguel J, Beksac M, Spicka I, Leleu X, Schjesvold F, Moreau P, Dimopoulos MA, Huang JS, Minarik J, Cavo M, Prince HM, Mace S, Corzo KP, Campana F, Le-Guennec S, Dubin F, Anderson KC; ICARIA-MM study group. Isatuximab plus pomalidomide and low-dose dexamethasone versus pomalidomide and low-dose dexamethasone in patients with relapsed and refractory multiple myeloma (ICARIA-MM): a randomised, multicentre, open-label, phase 3 study. Lancet. 2019 Dec 7;394(10214):2096-2107. doi: 10.1016/S0140-6736(19)32556-5. Epub 2019 Nov 14. PMID 31735560
- [Background] Richardson PG, Perrot A, San-Miguel J, Beksac M, Spicka I, Leleu X, Schjesvold F, Moreau P, Dimopoulos MA, Huang JS, Minarik J, Cavo M, Prince HM, Malinge L, Dubin F, van de Velde H, Anderson KC. Isatuximab plus pomalidomide and low-dose dexamethasone versus pomalidomide and low-dose dexamethasone in patients with relapsed and refractory multiple myeloma (ICARIA-MM): follow-up analysis of a randomised, phase 3 study. Lancet Oncol. 2022 Mar;23(3):416-427. doi: 10.1016/S1470-2045(22)00019-5. Epub 2022 Feb 10. PMID 35151415
- [Derived] Richardson PG, Perrot A, Miguel JS, Beksac M, Spicka I, Leleu X, Schjesvold F, Moreau P, Dimopoulos MA, Huang SY, Minarik J, Cavo M, Prince HM, Mace S, Zhang R, Dubin F, Morisse MC, Anderson KC. Isatuximab-pomalidomide-dexamethasone versus pomalidomide-dexamethasone in patients with relapsed and refractory multiple myeloma: final overall survival analysis. Haematologica. 2024 Jul 1;109(7):2239-2249. doi: 10.3324/haematol.2023.284325. PMID 38299578
- [Derived] Beksac M, Spicka I, Hajek R, Bringhen S, Jelinek T, Martin T, Mikala G, Moreau P, Symeonidis A, Rawlings AM, van de Velde H, Richardson PG. Evaluation of isatuximab in patients with soft-tissue plasmacytomas: An analysis from ICARIA-MM and IKEMA. Leuk Res. 2022 Nov;122:106948. doi: 10.1016/j.leukres.2022.106948. Epub 2022 Sep 6. PMID 36108425
- [Derived] Sunami K, Ikeda T, Huang SY, Wang MC, Koh Y, Min CK, Yeh SP, Matsumoto M, Uchiyama M, Iyama S, Shimazaki C, Lee JH, Kim K, Kaneko H, Kim JS, Lin TL, Campana F, Tada K, Iida S, Suzuki K; ICARIA-MM study group. Isatuximab-Pomalidomide-Dexamethasone Versus Pomalidomide-Dexamethasone in East Asian Patients With Relapsed/Refractory Multiple Myeloma: ICARIA-MM Subgroup Analysis. Clin Lymphoma Myeloma Leuk. 2022 Aug;22(8):e751-e761. doi: 10.1016/j.clml.2022.04.005. Epub 2022 Apr 8. PMID 35641409
- [Derived] Wilmoth J, Colson K, Dubin F, Kellam C. Isatuximab: Nursing Considerations for Use in the Treatment of Multiple Myeloma. Clin J Oncol Nurs. 2021 Dec 1;25(6):706-712. doi: 10.1188/21.CJON.706-712. PMID 34800109
- [Derived] Bringhen S, Pour L, Vorobyev V, Vural F, Warzocha K, Benboubker L, Koh Y, Maisnar V, Karlin L, Pavic M, Campana F, Le Guennec S, Menas F, van de Velde H, Richardson PG. Isatuximab plus pomalidomide and dexamethasone in patients with relapsed/refractory multiple myeloma according to prior lines of treatment and refractory status: ICARIA-MM subgroup analysis. Leuk Res. 2021 May;104:106576. doi: 10.1016/j.leukres.2021.106576. Epub 2021 Mar 29. PMID 33839618
- [Derived] Schjesvold FH, Richardson PG, Facon T, Alegre A, Spencer A, Jurczyszyn A, Sunami K, Frenzel L, Min CK, Guillonneau S, Lin PL, Le-Guennec S, Campana F, van de Velde H, Bensfia S, Bringhen S. Isatuximab plus pomalidomide and dexamethasone in elderly patients with relapsed/refractory multiple myeloma: ICARIA-MM subgroup analysis. Haematologica. 2021 Apr 1;106(4):1182-1187. doi: 10.3324/haematol.2020.253450. No abstract available. PMID 32586908

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 102 sites in 24 countries. A total of 387 participants were screened between 22 December 2016 and 01 February 2018. Out of which, 307 participants were randomized in 1:1 ratio to IPd (Isatuximab + Pomalidomide + Dexamethasone) and Pd (Pomalidomide + Dexamethasone) arms using an interactive response technology (IRT).
Pre-assignment Details: Randomization was stratified by age (less than [<] 75 years versus greater than and equal to [>=] 75 years) and number of previous lines of therapy (2 or 3 versus more than 3). "Reason for not completed" = "Reason for definitive treatment discontinuation."
Groups:
- Pd (Pomalidomide + Dexamethasone): Participants received pomalidomide 4 mg PO on Days 1 to 21 of each 28-day treatment cycle plus dexamethasone 40 mg (participants >= 75 years of age received 20 mg dexamethasone) PO on Days 1, 8, 15 and 22 of each 28-day treatment cycle until disease progression or unacceptable toxicity or participant's wish to discontinue study treatment, or any other reason, whichever comes first (maximum exposure: 306.6 weeks).
- IPd (Isatuximab + Pomalidomide + Dexamethasone): Participants received isatuximab 10 mg/kg IV infusion on Days 1, 8, 15, and 22 at Cycle 1, and then on Days 1 and 15 of subsequent cycles plus pomalidomide 4 mg PO on Days 1 to 21 of each 28-day treatment cycle and dexamethasone 40 mg (participants >= 75 years of age received 20 mg dexamethasone), PO or IV on Day 1, 8, 15, 22 of each 28-day treatment cycle until disease progression or unacceptable toxicity or participant's wish to discontinue study treatment, or any other reason, whichever comes first (maximum exposure: 311.0 weeks).
Period: Overall Study
Arm/Group | Pd (Pomalidomide + Dexamethasone) | IPd (Isatuximab + Pomalidomide + Dexamethasone)
Started | 153 | 154
Treated | 149 | 152
Completed | 0 | 0
Not Completed | 153 | 154
Not completed — Randomized and not treated | 4 | 2
Not completed — Adverse Event | 23 | 22
Not completed — Progressive disease | 118 | 107
Not completed — Poor compliance to protocol | 0 | 1
Not completed — Withdrawal by Subject | 6 | 8
Not completed — Physician's decision | 2 | 6
Not completed — Treatment extension study | 0 | 6
Not completed — Unconfirmed disease progression per investigator | 0 | 1
Not completed — Continue with therapy available commercially | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized population which included all participants with a signed informed consent and have been allocated a randomization number by the IRT, regardless of whether the participants was treated or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pd (Pomalidomide + Dexamethasone) | IPd (Isatuximab + Pomalidomide + Dexamethasone) | Total
Number analyzed (Participants) | 153 | 154 | 307
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (9.5) | 66.6 (9.1) | 65.9 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 65 | 148
  Male | 70 | 89 | 159
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 15 | 21 | 36
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 3 | 1 | 4
  White | 126 | 118 | 244
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 12 | 20

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS:time from date of randomization to date of first documentation of progressive disease (PD) determined by Independent Response Committee (IRC) or date of death from any cause, whichever comes first. If progression or death was not observed, participant was censored at date of last progression-free tumor assessment prior to study cut-off date. Analysis was performed by Kaplan-Meier method. PD as per International Myeloma Working Group (IMWG) criteria was defined as increase of >=25% from lowest confirmed value in any one of the following criteria: serum M-protein (the absolute increase must be >=0.5gram(g)/dL), serum M-protein increase >=1g/dL if lowest M component was >=5g/dL; urine M-component (absolute increase must be >=200mg/24hour), appearance of new lesion(s),>=50% increase from nadir in sum of the products of the maximal perpendicular diameters of measured lesions (SPD) of >1 lesion, or >=50% increase in the longest diameter of a previous lesion >1 centimeter in short axis.
Time Frame: From the date of randomization to the date of first documentation of progression, or the date of death from any cause, or initiation of further anti-myeloma treatment or data cut-off whichever comes first (maximum duration: 76.7 weeks)
Population: Analysis was performed on Intent-to-treat (ITT) population which included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Pd (Pomalidomide + Dexamethasone): Participants received pomalidomide 4 mg PO on Days 1 to 21 of each 28-day treatment cycle plus dexamethasone 40 mg (participants >= 75 years of age received 20 mg dexamethasone) PO on Days 1, 8, 15 and 22 of each 28-day treatment cycle until disease progression or unacceptable toxicity or participant's wish to discontinue study treatment, or any other reason, whichever comes first (maximum exposure: 73.7 weeks).
- IPd (Isatuximab + Pomalidomide + Dexamethasone): Participants received isatuximab 10 mg/kg IV infusion on Days 1, 8, 15, and 22 at Cycle 1, and then on Days 1 and 15 of subsequent cycles plus pomalidomide 4 mg PO on Days 1 to 21 of each 28-day treatment cycle and dexamethasone 40 mg (participants >= 75 years of age received 20 mg dexamethasone), PO or IV on Day 1, 8, 15, 22 of each 28-day treatment cycle until disease progression or unacceptable toxicity or participant's wish to discontinue study treatment, or any other reason, whichever comes first (maximum exposure: 76.7 weeks).
Arm/Group | Pd (Pomalidomide + Dexamethasone) | IPd (Isatuximab + Pomalidomide + Dexamethasone)
Number analyzed (Participants) | 153 | 154
months | 6.47 [4.468 to 8.279] | 11.53 [8.936 to 13.897]
Statistical Analysis 1: Comparison: Pd (Pomalidomide + Dexamethasone) vs IPd (Isatuximab + Pomalidomide + Dexamethasone); Confidence interval (CI) for Kaplan-Meier estimates were calculated with log-log transformation of survival function and methods of Brookmeyer and Crowley; Test type: Superiority — A closed test procedure was used to control the type I error rate meaning no further testing would be performed unless the significance level had been reached on PFS; p = 0.0005, Log Rank — One-sided p-value based on Stratified log-rank test. Threshold for statistical significance at 0.025; Stratification was based on age (<75 years versus >=75 years) and number of previous lines of therapy (2 or 3 versus >3) according to IRT; Hazard Ratio (HR) = 0.596, 95% CI 2-sided [0.436 to 0.814] — Stratification was based on age (<75 years versus >=75 years) and number of previous lines of therapy (2 or 3 versus >3) according to IRT

2. Secondary Outcome: Overall Response Rate (ORR): Percentage of Participants With Disease Response as Per Independent Response Committee (IRC)
Description: ORR (IMWG criteria): percentage of participants with stringent complete response(sCR), complete response (CR), very good partial response (VGPR), and partial response (PR) as best overall response, assessed by IRC. sCR:negative immunofixation on serum and urine,disappearance of any soft tissue plasmacytomas,<5% plasma cells in bone marrow aspirates plus normal free light chain(FLC)ratio(0.26-1.65), absence of clonal cells in bone marrow biopsy.CR:negative immunofixation on serum and urine,disappearance of any soft tissue plasmacytomas,<5% plasma cells in bone marrow aspirates.VGPR: serum and urine M-protein detectable by immunofixation, not on electrophoresis/,>=90% reduction in serum M-protein plus urine M-protein level <100mg/24h/,>=90% decrease in SPD compared to baseline in soft tissue plasmacytoma. PR: >=50% reduction of serum M-protein and reduction in 24h urinary M-protein by >=90%/<200mg/24h,if present at baseline,>=50% reduction in the size (SPD) of soft tissue plasmacytomas.
Time Frame: From the date of randomization to the date of first documentation of progression or initiation of further anti-myeloma treatment or data cut-off whichever comes first (maximum duration 76.7 weeks)
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Pd (Pomalidomide + Dexamethasone) | IPd (Isatuximab + Pomalidomide + Dexamethasone)
Number analyzed (Participants) | 153 | 154
percentage of participants | 35.3 | 60.4
Statistical Analysis 1: Comparison: Pd (Pomalidomide + Dexamethasone) vs IPd (Isatuximab + Pomalidomide + Dexamethasone); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for statistical significance at 0.025; One sided p-value was stratified based on age (<75 years versus >=75 years) and number of previous lines (2 or 3 versus >3) according to IRT

3. Secondary Outcome: Percentage of Participants With Best Overall Response (BOR) as Per Independent Response Committee
Description: BOR:best sequential response from start of treatment until disease progression, death, initiation of further anti-myeloma treatment/data cut-off, whichever comes first. Ordering of evaluations from best to worse was: sCR,CR,VGPR,PR, minimal response (MR), stable disease (SD), PD, and not evaluable.CR: negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas,<5% plasma cells in bone marrow aspirates. sCR:CR as defined previously plus normal FLC ratio (0.26 to 1.65), absence of clonal cells in bone marrow biopsy. VGPR: serum and urine M-protein detectable by immunofixation,>=90% reduction in serum M-protein plus urine M-protein level <100mg/24h,>=90% decrease in SPD compared to baseline in soft tissue plasmacytoma. PR: >=50% reduction of serum M-protein and reduction in 24h urinary M-protein by >=90%/<200mg/24h. MR:>=25% but <=49% reduction in serum M-protein and reduction in 24h urine M-protein by 50-89%. SD: Not meeting criteria for CR,VGPR,PR,MR/PD.
Time Frame: From the date of randomization until disease progression, or death, initiation of further anti-myeloma treatment or data cut-off whichever comes first (maximum duration 76.7 weeks)
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Pd (Pomalidomide + Dexamethasone) | IPd (Isatuximab + Pomalidomide + Dexamethasone)
Number analyzed (Participants) | 153 | 154
percentage of participants
  Stringent complete response | 0.7 | 0
  Complete response | 1.3 | 4.5
  Very good partial response | 6.5 | 27.3
  Partial response | 26.8 | 28.6
  Minimal response | 11.1 | 6.5
  Stable disease | 29.4 | 21.4
  Progressive Disease | 9.2 | 3.9
  Not evaluable | 10.5 | 4.5

4. Secondary Outcome: Percentage of Participants With Very Good Partial Response (VGPR) or Better as Per Independent Response Committee
Description: VGPR rate was defined as the percentage of participants achieving a VGPR or better as BOR. VGPR was defined as serum and urine M-protein detectable by immunofixation but not on electrophoresis or >=90% reduction in serum M-protein plus urine M-protein level <100 mg/24 h or >=90% decrease in the sum of maximal perpendicular diameter compared to baseline in soft tissue plasmacytoma. BOR was defined as the best sequential response, using the IRC's assessment of response, from the start of treatment until disease progression (provided that the progression is subsequently confirmed in case of progression requiring confirmation), death, initiation of further anti-myeloma treatment, or cut-off date, whichever occurs first. CR: negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas,<5% plasma cells in bone marrow aspirates.
Time Frame: From the date of randomization to the date of first documentation of progression, death, initiation of further anti-myeloma treatment, or data cut-off whichever comes first (maximum duration 76.7 weeks)
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Pd (Pomalidomide + Dexamethasone) | IPd (Isatuximab + Pomalidomide + Dexamethasone)
Number analyzed (Participants) | 153 | 154
percentage of participants | 8.5 | 31.8

5. Secondary Outcome: Clinical Benefit Rate (CBR): Percentage of Participants With Clinical Benefit as Per Independent Response Committee
Description: CBR was defined as the percentage of participants achieving a MR or better as BOR. MR was defined as >= 25% but <= 49% reduction in serum M-protein and reduction in 24h urine M-protein by 50-89%, which still exceed 200 mg/24h; if present at baseline, >=50% reduction in size (SPD) of soft tissue plasmacytomas was also required. BOR was defined as the best sequential response, using the IRC's assessment of response, from the start of treatment until disease progression (provided that the progression is subsequently confirmed in case of progression requiring confirmation), death, initiation of further anti-myeloma treatment, or cut-off date, whichever occurs first.
Time Frame: From the date of randomization to the date of first documentation of progression, death, initiation of further anti-myeloma treatment or data cut-off whichever comes first (maximum duration 76.7 weeks)
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Pd (Pomalidomide + Dexamethasone) | IPd (Isatuximab + Pomalidomide + Dexamethasone)
Number analyzed (Participants) | 153 | 154
percentage of participants | 46.4 | 66.9

6. Secondary Outcome: Overall Survival (OS): Final Analysis
Description: OS was defined as the time from the date of randomization to death from any cause. In the absence of confirmation of death, survival time was censored at the last date participant was known to be alive or at the cut-off date, whichever comes first. This pre-specified final analysis was performed when the 220 OS events were met.
Time Frame: From the date of randomization to date of death from any cause or data cut-off date, whichever was earlier (maximum duration 245.6 weeks)
Population: Analysis was performed on ITT population.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Pd (Pomalidomide + Dexamethasone): Participants received pomalidomide 4 mg PO on Days 1 to 21 of each 28-day treatment cycle plus dexamethasone 40 mg (participants >= 75 years of age received 20 mg dexamethasone) PO on Days 1, 8, 15 and 22 of each 28-day treatment cycle until disease progression or unacceptable toxicity or participant's wish to discontinue study treatment, or any other reason, whichever comes first (maximum exposure: 241.6 weeks).
- IPd (Isatuximab + Pomalidomide + Dexamethasone): Participants received isatuximab 10 mg/kg IV infusion on Days 1, 8, 15, and 22 at Cycle 1, and then on Days 1 and 15 of subsequent cycles plus pomalidomide 4 mg PO on Days 1 to 21 of each 28-day treatment cycle and dexamethasone 40 mg (participants >= 75 years of age received 20 mg dexamethasone), PO or IV on Day 1, 8, 15, 22 of each 28-day treatment cycle until disease progression or unacceptable toxicity or participant's wish to discontinue study treatment, or any other reason, whichever comes first (maximum exposure: 245.6 weeks).
Arm/Group | Pd (Pomalidomide + Dexamethasone) | IPd (Isatuximab + Pomalidomide + Dexamethasone)
Number analyzed (Participants) | 153 | 154
months | 17.71 [14.390 to 26.218] | 24.57 [20.304 to 31.310]
Statistical Analysis 1: Comparison: Pd (Pomalidomide + Dexamethasone) vs IPd (Isatuximab + Pomalidomide + Dexamethasone); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0319, Log Rank — One-sided significance level was 0.02 using the O'Brien-Fleming alpha spending function; Stratified on age (<75 years versus >=75 years) and number of previous lines of therapy (2 or 3 versus > 3) according to IRT; Hazard Ratio (HR) = 0.776, 95% CI 2-sided [0.594 to 1.015] — Stratified on age (<75 years versus >=75 years) and number of previous lines of therapy (2 or 3 versus > 3) according to IRT

7. Secondary Outcome: Time to Progression (TTP) as Per Independent Response Committee
Description: TTP was defined as time from randomization to the date of first documentation of PD, as determined by the IRC. As per IMWG criteria, PD was defined for participants with increase of >= 25% from lowest confirmed value in any one of the following criteria: serum M-protein (the absolute increase must be >= 0.5 g/dL), serum M-protein increase >=1 g/dL if the lowest M component was >=5 g/dL; urine M-component (the absolute increase must be >=200 mg/24hour), appearance of new lesion(s), >=50% increase from nadir in SPD of >1 lesion, or >=50% increase in the longest diameter of a previous lesion >1 centimeter in short axis.
Time Frame: From the date of randomization to the date of first documentation of progression, or initiation of further anti-myeloma treatment or data cut-off whichever comes first (maximum duration 76.7 weeks)
Population: Analysis was performed on ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pd (Pomalidomide + Dexamethasone) | IPd (Isatuximab + Pomalidomide + Dexamethasone)
Number analyzed (Participants) | 153 | 154
months | 7.75 [5.027 to 9.758] | 12.71 [11.203 to 15.211]

8. Secondary Outcome: Progression Free Survival in High Risk Cytogenetic Population
Description: PFS in high risk cytogenetic population was defined as PFS in subgroup of participants carrying high risk cytogenetic changes including del(17p), translocation (t)(4;14) or translocation t(14;16) assessed by fluorescence in situ hybridization (FISH). PFS was defined as the time from date of randomization to date of first documentation of PD (determined by IRC) or date of death from any cause, whichever comes first. PD defined as per IMWG criteria as: increase of >=25% from lowest confirmed value in any one of following criteria: serum M-protein (absolute increase must be >=0.5 g/dL), serum M-protein increase >=1 g/dL if lowest M component was >=5 g/dL; urine M-component (absolute increase must be >=200 mg/24hour), appearance of new lesion(s), >=50% increase from nadir in SPD of >1 lesion, or >=50% increase in the longest diameter of previous lesion >1 centimeter (cm) in short axis.
Time Frame: From the date of randomization to the date of first documentation of progression, or the date of death from any cause, or initiation of further anti-myeloma treatment or data cut-off whichever comes first (maximum duration 76.7 weeks)
Population: Analysis was performed in high-risk cytogenetic population which included participants carrying del (17p), t(4;14) or t(14;16) in each arm.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pd (Pomalidomide + Dexamethasone) | IPd (Isatuximab + Pomalidomide + Dexamethasone)
Number analyzed (Participants) | 36 | 25
months | 3.745 [2.793 to 7.885] | 7.491 [2.628 to NA] — Due to smaller number of participants with an event, 95% CI could not be calculated.

9. Secondary Outcome: Duration of Response (DOR) as Per Independent Response Committee
Description: DOR:time from date of first IRC determined response(PR or better) to date of first IRC-PD or death, whichever occurred first.DOR was determined only for participants who had achieved a response of PR or better based on disease assessment by IRC.If progression or death was not observed,participant was censored at date of participants last progression-free tumor assessment prior to initiation of further anti-myeloma treatment(if any)and study cut-off date. PD(IMWG criteria):increase of >=25% from lowest confirmed value in any one of following criteria: serum M-protein (absolute increase must be >=0.5 g/dL), serum M-protein increase >=1g/dL if lowest M component was >=5g/dL;urine M-component (absolute increase must be >=200mg/24 hour),appearance of new lesion(s), >=50% increase from nadir in SPD of >1 lesion,or >=50% increase in the longest diameter of a previous lesion >1 cm in short axis. PR:>=50% reduction of serum M-protein and reduction in 24h urinary M-protein by >=90%/<200mg/24h.
Time Frame: From the date of the first IRC determined response to the date of first IRC progression or death, whichever occurred first (maximum duration 76.7 weeks)
Population: Analysis was performed on responders in ITT population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pd (Pomalidomide + Dexamethasone) | IPd (Isatuximab + Pomalidomide + Dexamethasone)
Number analyzed (Participants) | 54 | 93
months | 11.07 [8.542 to NA] — Due to smaller number of participants with an event, 95% CI could not be calculated. | 13.27 [10.612 to NA] — Due to smaller number of participants with an event, 95% CI could not be calculated.

10. Secondary Outcome: Time to First Response (TT1R) as Per Independent Response Committee
Description: TT1R was defined as the time from randomization to the date of first IRC determined response (PR or better) that is subsequently confirmed. PR was defined as >=50% reduction of serum M-protein and reduction in 24 hours urinary M-protein by >=90% or to <200 mg/24 h. In addition to the above listed criteria, if present at baseline, a >=50% reduction in the size (SPD) of soft tissue plasmacytomas was also required.
Time Frame: From the date of randomization to the date of first IRC determined response, or death or data cut-off whichever comes first (maximum duration 76.7 weeks)
Population: Analysis was performed on ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pd (Pomalidomide + Dexamethasone) | IPd (Isatuximab + Pomalidomide + Dexamethasone)
Number analyzed (Participants) | 153 | 154
months | 3.02 [2.825 to 5.060] | 1.94 [1.314 to 2.004]

11. Secondary Outcome: Time to Best Response (TTBR) as Per Independent Response Committee
Description: TTBR was defined as the time from randomization to the date of first occurrence of IRC determined BOR (PR or better) that was subsequently confirmed. PR was defined as >=50% reduction of serum M-protein and reduction in 24 hours urinary M-protein by >=90% or to <200 mg/24 h. In addition to the above listed criteria, if present at baseline, a >=50% reduction in the size (SPD) of soft tissue plasmacytomas was also required. BOR was defined as the best sequential response, using the IRC's assessment of response, from the start of treatment until disease progression (provided that the progression is subsequently confirmed in case of progression requiring confirmation), death, initiation of further anti-myeloma treatment, or cut-off date, whichever occurs first.
Time Frame: From the date of randomization to date of first occurrence of IRC determined best overall response or data cut-off whichever comes first (maximum duration 76.7 weeks)
Population: Analysis was performed on ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pd (Pomalidomide + Dexamethasone) | IPd (Isatuximab + Pomalidomide + Dexamethasone)
Number analyzed (Participants) | 153 | 154
months | 5.06 [3.778 to 7.885] | 4.30 [2.891 to 5.125]

12. Secondary Outcome: Number of Participants With Minimal Residual Disease (MRD)
Description: MRD was assessed by next-generation sequencing in bone marrow samples from participants who achieved CR, to determine the depth of response at the molecular level. IMWG criteria for CR: Negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas, and <5% plasma cells in bone marrow aspirates. MRD was classified as positive or negative at the minimum sensitivity of 1 in 10^5 nucleated cells. MRD negativity was defined as the absence of the dominant clonotype sequence(s) identified in the bone marrow aspirate collected at screening. MRD positivity was defined as the presence of the dominant clonotype sequence(s) identified in the bone marrow aspirate collected at screening.
Time Frame: Up to 76.7 weeks
Population: Analysis was performed on ITT population who were evaluable for MRD.
Measure: Count of Participants; unit: Participants
Arm/Group | Pd (Pomalidomide + Dexamethasone) | IPd (Isatuximab + Pomalidomide + Dexamethasone)
Number analyzed (Participants) | 2 | 14
Participants
  MRD negative:1 in 10^4 | 0 | 10
  MRD negative:1 in 10^5 | 0 | 8
  MRD negative:1 in 10^6 | 0 | 2
  MRD positive:1 in 10^4 | 2 | 4
  MRD positive:1 in 10^5 | 2 | 6
  MRD positive:1 in 10^6 | 2 | 9

13. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Adverse Event (AE) was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily had a causal relationship with the treatment. TEAEs were defined as AEs that developed, worsened (according to the Investigator opinion), or became serious during the treatment period (time from the first dose of study treatments up to 30 days after last dose of study treatments). An SAE is any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a medically important event.
Time Frame: From randomization up to 30 days after last dose of study drug (maximum duration up to 241.6 weeks for Pd arm and 245.6 weeks for IPd arm)
Population: Analysis was performed on safety population which included all participants from the ITT population who received at least one dose or a part of a dose of the study treatments.
Measure: Count of Participants; unit: Participants
Arm/Group | Pd (Pomalidomide + Dexamethasone) | IPd (Isatuximab + Pomalidomide + Dexamethasone)
Number analyzed (Participants) | 149 | 152
Participants
  Any TEAE | 146 | 151
  Any treatment emergent SAE | 91 | 112
  Any TEAE leading to treatment discontinuation | 22 | 19

14. Secondary Outcome: Pharmacokinetics (PK) Parameter: Plasma Concentration of Isatuximab at End of Infusion (CEOI)
Description: CEOI was defined as the plasma concentration at end of infusion.
Time Frame: End of infusion on Cycle(C)1 Day(D)1 and Cycle1 Day 15; Cycle 2 Day 1; and Cycle 4 Day 1
Population: Analysis was performed on PK population which included participants who received at least 1 dose of Isatuximab, with data for at least 1 PK parameter available. Here, 'Number analyzed' = participants with available data for each specified category. Data for this outcome measure (OM) was not planned to be collected and analyzed for Pd arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (mcg/mL)
Arm/Group | IPd (Isatuximab + Pomalidomide + Dexamethasone)
Number analyzed (Participants) | 149
microgram per milliliter (mcg/mL)
  End of infusion: C1D1: number analyzed (Participants) | 141
  End of infusion: C1D1 | 163.05 (34.528)
  End of infusion: C1D15: number analyzed (Participants) | 120
  End of infusion: C1D15 | 269.20 (32.622)
  End of infusion: C2D1: number analyzed (Participants) | 134
  End of infusion: C2D1 | 299.85 (35.921)
  End of infusion: C4D1: number analyzed (Participants) | 117
  End of infusion: C4D1 | 279.31 (47.555)

15. Secondary Outcome: Pharmacokinetic Parameter: Accumulation Ratio of Isatuximab at Concentration at the End of Infusion (CEOI)
Description: Accumulation Ratio was defined as the ratio of CEOI of Cycle 2 Day 1 versus Cycle 1 Day 1 and Cycle 4 Day 1 versus Cycle 1 Day 1, where CEOI was the plasma concentration at the end of infusion.
Time Frame: End of infusion on Cycle 1 Day 1, Cycle 2 Day 1, and Cycle 4 Day 1
Population: Analysis was performed on PK population. Here, 'Number analyzed' = participants with available data for each specified category. Data for this OM was not planned to be collected and analyzed for Pd arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | IPd (Isatuximab + Pomalidomide + Dexamethasone)
Number analyzed (Participants) | 149
ratio
  C2D1 versus C1D1: number analyzed (Participants) | 130
  C2D1 versus C1D1 | 1.860 (170.9185)
  C4D1 versus C1D1: number analyzed (Participants) | 112
  C4D1 versus C1D1 | 1.777 (224.2542)

16. Secondary Outcome: Pharmacokinetic Parameter: Plasma Concentration of Isatuximab at 1 Hour After End of Infusion (CEOI+1 Hour)
Description: CEOI+1 hour was defined as the plasma concentration of isatuximab at 1 hour after end of infusion.
Time Frame: Cycle 1:1 hour after End of Infusion on Day 1; Cycle 4:1 hour after End of Infusion on Day 1
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | IPd (Isatuximab + Pomalidomide + Dexamethasone)
Number analyzed (Participants) | 149
mcg/mL
  C1D1: number analyzed (Participants) | 140
  C1D1 | 171.55 (38.299)
  C4D1: number analyzed (Participants) | 114
  C4D1 | 294.96 (57.331)

17. Secondary Outcome: PK Parameter: Plasma Concentration of Isatuximab at Ctrough
Description: Trough Concentration (Ctrough) is the concentration prior to study drug administration.
Time Frame: Pre-infusion on C1D1, C1D8, C1D15, C1D22, C2D1, C2D15, C3D1, C3D15, C4D1, C4D15, C5D1, C6D1, C7D1, C8D1, C9D1, C10D1, C11D1, C12D1, C13D1, C14D1, C15D1, C16D1, C17D1, C18D1, C19D1, C20D1; End of treatment (EOT [30 days after last drug administration])
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | IPd (Isatuximab + Pomalidomide + Dexamethasone)
Number analyzed (Participants) | 149
mcg/mL
  C1D1: number analyzed (Participants) | 144
  C1D1 | 0.00 (1194.973)
  C1D8: number analyzed (Participants) | 135
  C1D8 | 31.49 (53.602)
  C1D15: number analyzed (Participants) | 126
  C1D15 | 57.89 (54.764)
  C1D22: number analyzed (Participants) | 126
  C1D22 | 84.82 (57.666)
  C2D1: number analyzed (Participants) | 138
  C2D1 | 89.09 (60.155)
  C2D15: number analyzed (Participants) | 121
  C2D15 | 89.35 (61.167)
  C3D1: number analyzed (Participants) | 131
  C3D1 | 64.15 (76.469)
  C3D15: number analyzed (Participants) | 109
  C3D15 | 91.73 (78.406)
  C4D1: number analyzed (Participants) | 118
  C4D1 | 86.05 (70.062)
  C4D15: number analyzed (Participants) | 108
  C4D15 | 105.42 (68.035)
  C5D1: number analyzed (Participants) | 108
  C5D1 | 106.08 (65.275)
  C6D1: number analyzed (Participants) | 107
  C6D1 | 111.33 (64.985)
  C7D1: number analyzed (Participants) | 96
  C7D1 | 134.14 (60.017)
  C8D1: number analyzed (Participants) | 86
  C8D1 | 146.15 (55.946)
  C9D1: number analyzed (Participants) | 82
  C9D1 | 162.84 (65.193)
  C10D1: number analyzed (Participants) | 73
  C10D1 | 145.86 (60.719)
  C11D1: number analyzed (Participants) | 71
  C11D1 | 169.39 (56.078)
  C12D1: number analyzed (Participants) | 63
  C12D1 | 182.32 (56.814)
  C13D1: number analyzed (Participants) | 49
  C13D1 | 215.85 (54.667)
  C14D1: number analyzed (Participants) | 35
  C14D1 | 214.88 (55.172)
  C15D1: number analyzed (Participants) | 24
  C15D1 | 253.61 (58.885)
  C16D1: number analyzed (Participants) | 19
  C16D1 | 206.60 (50.965)
  C17D1: number analyzed (Participants) | 13
  C17D1 | 242.79 (45.364)
  C18D1: number analyzed (Participants) | 8
  C18D1 | 216.70 (58.273)
  C19D1: number analyzed (Participants) | 5
  C19D1 | 240.36 (42.099)
  C20D1: number analyzed (Participants) | 1
  C20D1 | 164.07
  EOT: number analyzed (Participants) | 60
  EOT | 9.51 (136.883)

18. Secondary Outcome: PK Parameter: Accumulation Ratio of Isatuximab at Trough Concentration (Ctrough)
Description: Accumulation Ratio was defined as the ratio of Ctrough of Cycle 2 Day 1 versus Cycle 1 Day 8 and Cycle 4 Day 1 versus Cycle 1 Day 8, where Ctrough is the concentration prior to study drug administration.
Time Frame: Pre-infusion on Cycle 1 Day 8, Cycle 2 Day 1, and Cycle 4 Day 1
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | IPd (Isatuximab + Pomalidomide + Dexamethasone)
Number analyzed (Participants) | 149
ratio
  C2D1 versus C1D8: number analyzed (Participants) | 125
  C2D1 versus C1D8 | 2.689 (734.5547)
  C4D1 versus C1D8: number analyzed (Participants) | 108
  C4D1 versus C1D8 | 2.620 (645.4171)

19. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA)
Description: ADA were categorized as: pre-existing, treatment induced and treatment boosted response. Pre-existing ADA was defined as ADA that were present in samples drawn during the pretreatment period (i.e., before the first isatuximab administration). Treatment-induced ADA was defined as ADA that developed at any time during the ADA on-study observation period in participants without preexisting ADA, including participants without pretreatment samples. Treatment boosted ADA was defined as pre-existing ADA that increased at least 2 titer steps between pre-treatment and post-treatment.
Time Frame: From randomization up to 60 days after last dose of study drug (maximum duration 76.7 weeks)
Population: Analysis was performed on ADA evaluable population which included participants who received at least one dose of study drug from the IPd arm with at least one ADA assessment during the ADA on-study observation period with a reportable result. Data for this OM was not planned to be collected and analyzed for Pd arm.
Measure: Count of Participants; unit: Participants
Arm/Group | IPd (Isatuximab + Pomalidomide + Dexamethasone)
Number analyzed (Participants) | 151
Participants
  Pre-existing ADA | 0
  Treatment induced ADA | 0
  Treatment boosted ADA | 0

20. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Cancer Specific Questionnaire With 30 Items (EORTC QLQ-C30): Global Health Status (GHS)/Quality of Life (QOL) Score
Description: EORTC-Quality of Life Questionnaire (QLQ)-C30 is a cancer-specific instrument with 30 questions for evaluation of new chemotherapy and provides an assessment of participant reported outcome dimensions. EORTC QLQ-C30 included GHS/ QOL, functional scales (physical, role, cognitive, emotional, social), symptom scales (fatigue, pain, nausea/vomiting), and 6 single items (dyspnea, appetite loss, insomnia, constipation, diarrhea, financial difficulties). Most questions from QLQ-C30 were a 4-point scale (1/Not at All to 4/Very Much), except Items 29-30, which comprise GHS scale and were a 7-point scale (1/Very Poor to 7/Excellent). Answers were converted into grading scale, with values between 0 and 100. A high score represented a favorable outcome with a best quality of life for participant.
Time Frame: Baseline, Day 1 of each cycle (Cycle 3, Cycle 6, Cycle 9, and Cycle 17)
Population: Analysis was performed on safety population evaluable for global health status. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pd (Pomalidomide + Dexamethasone) | IPd (Isatuximab + Pomalidomide + Dexamethasone)
Number analyzed (Participants) | 134 | 139
score on a scale
  Baseline: number analyzed (Participants) | 134 | 137
  Baseline | 61.19 (20.64) | 60.10 (20.02)
  Day 1: Cycle 3: number analyzed (Participants) | 109 | 123
  Day 1: Cycle 3 | -1.45 (21.03) | -1.22 (22.42)
  Day 1: Cycle 6: number analyzed (Participants) | 69 | 102
  Day 1: Cycle 6 | -0.12 (22.26) | -0.16 (18.28)
  Day 1: Cycle 9: number analyzed (Participants) | 55 | 82
  Day 1: Cycle 9 | 1.06 (19.97) | 0.41 (20.99)
  Day 1: Cycle 17: number analyzed (Participants) | 10 | 13
  Day 1: Cycle 17 | -9.17 (24.36) | -1.92 (19.29)

21. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Multiple Myeloma Specific Module With 20 Items (EORTC QLQ-MY20): Disease Symptoms Domain Score
Description: EORTC QLQ-MY20 is a validated questionnaire to assess the overall quality of life in participants with multiple myeloma. Disease symptoms domain is one of the four domain scores. Disease symptoms domain score used 4-point scale (1 'Not at All' to 4 'Very Much'). Scores are averaged, and transformed to 0 -100 scale, where higher scores = more symptoms and lower health-related quality of life (HRQL) and lower score = less symptoms and more HRQL
Time Frame: Baseline, Day 1 of each cycle (Cycle 3, Cycle 6, Cycle 9, and Cycle 17)
Population: Analysis was performed on safety population evaluable for disease symptoms. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pd (Pomalidomide + Dexamethasone) | IPd (Isatuximab + Pomalidomide + Dexamethasone)
Number analyzed (Participants) | 130 | 137
score on a scale
  Baseline: number analyzed (Participants) | 130 | 135
  Baseline | 24.91 (20.67) | 24.12 (20.54)
  Day 1: Cycle 3: number analyzed (Participants) | 107 | 121
  Day 1: Cycle 3 | -3.79 (16.09) | -2.07 (17.51)
  Day 1: Cycle 6: number analyzed (Participants) | 68 | 101
  Day 1: Cycle 6 | -4.08 (17.95) | -3.30 (16.01)
  Day 1: Cycle 9: number analyzed (Participants) | 55 | 81
  Day 1: Cycle 9 | -2.83 (15.04) | -4.66 (13.73)
  Day 1: Cycle 17: number analyzed (Participants) | 10 | 13
  Day 1: Cycle 17 | -3.33 (15.54) | 0.00 (21.40)

22. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Multiple Myeloma Specific Module With 20 Items (EORTC QLQ-MY20): Side Effects of Treatment Domain Score
Description: EORTC QLQ-MY20 is a validated questionnaire to assess the overall quality of life in participants with multiple myeloma. Side effects of treatment domain is one of the four domain scores. Side effects of treatment domain score used 4-point scale (1 'Not at All' to 4 'Very Much'). Scores are averaged, and transformed to 0-100 scale, where higher scores = more side effects and lower HRQL and lower scores = less side effects and better HRQL.
Time Frame: Baseline, Day 1 of each cycle (Cycle 3, Cycle 6, Cycle 9, and Cycle 17)
Population: Analysis was performed on safety population evaluable for side effects of treatment. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pd (Pomalidomide + Dexamethasone) | IPd (Isatuximab + Pomalidomide + Dexamethasone)
Number analyzed (Participants) | 130 | 137
score on a scale
  Baseline: number analyzed (Participants) | 130 | 135
  Baseline | 17.49 (15.25) | 15.60 (11.63)
  Day 1: Cycle 3: number analyzed (Participants) | 107 | 121
  Day 1: Cycle 3 | 1.69 (11.54) | 2.61 (13.39)
  Day 1: Cycle 6: number analyzed (Participants) | 68 | 101
  Day 1: Cycle 6 | -0.13 (15.10) | 2.11 (11.78)
  Day 1: Cycle 9: number analyzed (Participants) | 55 | 81
  Day 1: Cycle 9 | 1.43 (14.66) | 3.14 (11.88)
  Day 1: Cycle 17: number analyzed (Participants) | 10 | 13
  Day 1: Cycle 17 | -2.93 (15.94) | 3.02 (15.72)

23. Secondary Outcome: Change From Baseline in European Quality of Life Working Group Health Status Measure 5 Dimensions (5D), 5 Levels (5L) (EQ-5D-5L) Score: Health State Utility Index Value
Description: The EQ-5D-5L is a standardized measure of health status that provides a general assessment of health and wellbeing. The EQ-5D descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has a 5-level response: no problems, slight problems, moderate problems, severe problems, and extreme problems. Response options are measured with a 5-point Likert scale (for the 5L version). The 5D-5L systems are converted into a single index utility score between 0 to 1, where higher score indicates a better health state and lower score indicate worse health state.
Time Frame: Baseline, Day 1 of each cycle (Cycle 3, Cycle 6, Cycle 9, and Cycle 17)
Population: Analysis was performed on safety population evaluable for health state utility index. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pd (Pomalidomide + Dexamethasone) | IPd (Isatuximab + Pomalidomide + Dexamethasone)
Number analyzed (Participants) | 134 | 140
score on a scale
  Baseline: number analyzed (Participants) | 134 | 138
  Baseline | 0.70 (0.24) | 0.71 (0.21)
  Day 1: Cycle 3: number analyzed (Participants) | 109 | 125
  Day 1: Cycle 3 | -0.01 (0.22) | -0.01 (0.22)
  Day 1: Cycle 6: number analyzed (Participants) | 69 | 101
  Day 1: Cycle 6 | 0.02 (0.22) | -0.00 (0.20)
  Day 1: Cycle 9: number analyzed (Participants) | 55 | 82
  Day 1: Cycle 9 | -0.03 (0.27) | -0.01 (0.15)
  Day 1: Cycle 17: number analyzed (Participants) | 10 | 13
  Day 1: Cycle 17 | -0.02 (0.19) | -0.01 (0.23)

24. Secondary Outcome: Change From Baseline in European Quality of Life Working Group Health Status Measure 5 Dimensions, 5 Levels (EQ-5D-5L) Score: Visual Analogic Scale (VAS)
Description: EQ-5D-5L is a standardized, participant-rated questionnaire to assess health-related quality of life. The EQ-5D-5L includes 2 components: the EQ-5D-5L health state utility index (descriptive system) and the EQ-5D-5L Visual Analog Scale. The Visual Analogue Scale is designed to rate the participant's current health state on a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state.
Time Frame: Baseline, Day 1 of each cycle (Cycle 3, Cycle 6, Cycle 9, and Cycle 17)
Population: Analysis was performed on safety population evaluable for visual analogue scale. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Pd (Pomalidomide + Dexamethasone) | IPd (Isatuximab + Pomalidomide + Dexamethasone)
Number analyzed (Participants) | 134 | 140
centimeter
  Baseline: number analyzed (Participants) | 134 | 138
  Baseline | 65.38 (19.31) | 66.62 (19.32)
  Day 1: Cycle 3: number analyzed (Participants) | 109 | 125
  Day 1: Cycle 3 | 0.26 (17.37) | 0.92 (19.41)
  Day 1: Cycle 6: number analyzed (Participants) | 69 | 101
  Day 1: Cycle 6 | 2.49 (18.83) | 1.19 (17.70)
  Day 1: Cycle 9: number analyzed (Participants) | 55 | 82
  Day 1: Cycle 9 | 4.42 (19.78) | 1.96 (16.60)
  Day 1: Cycle 17: number analyzed (Participants) | 10 | 13
  Day 1: Cycle 17 | -1.70 (12.39) | -3.00 (12.58)

ADVERSE EVENTS:
Time Frame: AE data was collected from the time of first dose of study drug administration up to 30 days following the last administration of study treatment (maximum duration up to 306.6 weeks for Pd arm and 311.0 weeks for IPd arm). Per participant, the deaths were collected up to a maximum duration of approximately 72.38 months.
Description: All-Cause Mortality was assessed for all randomized participants, Serious and Other Adverse Events were collected for safety population only.
Arm/Group | Pd (Pomalidomide + Dexamethasone) | IPd (Isatuximab + Pomalidomide + Dexamethasone)
All-Cause Mortality (participants affected / at risk) | 115/153 | 110/154
Serious Adverse Events (participants affected / at risk) | 91/149 | 112/152
Other Adverse Events (participants affected / at risk) | 139/149 | 145/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pd (Pomalidomide + Dexamethasone) (N=149) | IPd (Isatuximab + Pomalidomide + Dexamethasone) (N=152)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1)
Atypical Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Bronchiolitis (Infections and infestations) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 7 (8)
Covid-19 (Infections and infestations) | 2 (2) | 0 (0)
Covid-19 Pneumonia (Infections and infestations) | 3 (3) | 2 (2)
Candida Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis Staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Coronavirus Infection (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus Gastrointestinal Infection (Infections and infestations) | 1 (1) | 0 (0)
Device Related Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 2 (2)
Ear, Nose And Throat Infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis Enteroviral (Infections and infestations) | 0 (0) | 1 (1)
Haemophilus Infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes Zoster Disseminated (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 4 (4)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Lower Respiratory Tract Infection (Infections and infestations) | 3 (3) | 7 (8)
Lymphangitis (Infections and infestations) | 0 (0) | 1 (1)
Medical Device Site Infection (Infections and infestations) | 0 (0) | 1 (1)
Meningitis Cryptococcal (Infections and infestations) | 0 (0) | 1 (1)
Meningitis Listeria (Infections and infestations) | 0 (0) | 1 (1)
Neurological Infection (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Periorbital Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 5 (5) | 4 (4)
Pneumonia (Infections and infestations) | 31 (33) | 35 (51)
Pneumonia Bacterial (Infections and infestations) | 1 (1) | 5 (6)
Pneumonia Fungal (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia Haemophilus (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia Influenzal (Infections and infestations) | 2 (2) | 2 (2)
Pneumonia Pneumococcal (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia Streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Viral (Infections and infestations) | 0 (0) | 3 (3)
Postoperative Wound Infection (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonal Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonas Infection (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis Acute (Infections and infestations) | 1 (1) | 0 (0)
Pyoderma (Infections and infestations) | 0 (0) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 2 (2) | 2 (2)
Sepsis (Infections and infestations) | 2 (2) | 4 (4)
Septic Shock (Infections and infestations) | 4 (4) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin Infection (Infections and infestations) | 0 (0) | 1 (1)
Soft Tissue Infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Systemic Candida (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 5 (5) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 7 (8)
Varicella (Infections and infestations) | 0 (0) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lip Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lip Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Metastatic Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (5)
Tumour Associated Fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (4)
Febrile Neutropenia (Blood and lymphatic system disorders) | 5 (5) | 10 (12)
Hyperviscosity Syndrome (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 5 (5)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Splenic Infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (4) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic Disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acute Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional State (Psychiatric disorders) | 1 (1) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Basal Ganglia Infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cauda Equina Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar Infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Depressed Level Of Consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage Intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial Aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Spinal Subdural Haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 4 (4)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 2 (2)
Vith Nerve Paresis (Nervous system disorders) | 0 (0) | 1 (1)
Vocal Cord Paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 2 (2)
Retinal Detachment (Eye disorders) | 1 (1) | 0 (0)
Vision Blurred (Eye disorders) | 1 (1) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 2 (2)
Angina Pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Angina Unstable (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia Supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 3 (4)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure Chronic (Cardiac disorders) | 0 (0) | 1 (1)
Diastolic Dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 3 (3)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Orthostatic Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (2)
Colitis Ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diverticular Perforation (Gastrointestinal disorders) | 0 (0) | 2 (3)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large Intestine Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bile Duct Stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic Foot (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis Of Jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporotic Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (7)
Soft Tissue Necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 6 (8) | 6 (6)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Aneurysm (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 3 (4) | 1 (1)
Renal Impairment (Renal and urinary disorders) | 0 (0) | 2 (2)
Pelvic Pain (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 2 (2)
Disease Progression (General disorders) | 8 (8) | 9 (9)
General Physical Health Deterioration (General disorders) | 3 (3) | 1 (1)
Influenza Like Illness (General disorders) | 0 (0) | 1 (1)
Multiple Organ Dysfunction Syndrome (General disorders) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1)
Peripheral Swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 5 (5)
Sudden Death (General disorders) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1)
Hepatic Enzyme Increased (Investigations) | 0 (0) | 1 (1)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 (1) | 6 (6)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pd (Pomalidomide + Dexamethasone) (N=149) | IPd (Isatuximab + Pomalidomide + Dexamethasone) (N=152)
Bronchitis (Infections and infestations) | 16 (29) | 37 (65)
Influenza (Infections and infestations) | 6 (7) | 8 (9)
Nasopharyngitis (Infections and infestations) | 10 (13) | 23 (44)
Oral Herpes (Infections and infestations) | 3 (3) | 9 (18)
Pneumonia (Infections and infestations) | 10 (10) | 18 (29)
Upper Respiratory Tract Infection (Infections and infestations) | 28 (51) | 53 (121)
Urinary Tract Infection (Infections and infestations) | 13 (15) | 15 (21)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 8 (10)
Neutropenia (Blood and lymphatic system disorders) | 52 (96) | 77 (192)
Thrombocytopenia (Blood and lymphatic system disorders) | 17 (19) | 19 (27)
Decreased Appetite (Metabolism and nutrition disorders) | 8 (9) | 17 (23)
Insomnia (Psychiatric disorders) | 14 (17) | 15 (17)
Dizziness (Nervous system disorders) | 5 (5) | 10 (11)
Headache (Nervous system disorders) | 9 (9) | 16 (19)
Peripheral Sensory Neuropathy (Nervous system disorders) | 11 (11) | 18 (20)
Tremor (Nervous system disorders) | 7 (7) | 13 (14)
Cataract (Eye disorders) | 11 (11) | 13 (14)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 8 (11)
Hypertension (Vascular disorders) | 7 (9) | 11 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (15) | 14 (22)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 23 (33)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 12 (15)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (12)
Abdominal Pain (Gastrointestinal disorders) | 6 (7) | 8 (8)
Constipation (Gastrointestinal disorders) | 30 (35) | 27 (37)
Diarrhoea (Gastrointestinal disorders) | 32 (44) | 49 (86)
Nausea (Gastrointestinal disorders) | 14 (14) | 24 (27)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 10 (14)
Vomiting (Gastrointestinal disorders) | 6 (6) | 20 (22)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (12) | 9 (9)
Rash (Skin and subcutaneous tissue disorders) | 8 (8) | 11 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (18) | 19 (22)
Back Pain (Musculoskeletal and connective tissue disorders) | 24 (25) | 29 (32)
Bone Pain (Musculoskeletal and connective tissue disorders) | 13 (14) | 11 (13)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 17 (20) | 18 (19)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 8 (8) | 13 (14)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 15 (16)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 12 (14)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 12 (12)
Asthenia (General disorders) | 29 (36) | 23 (37)
Fatigue (General disorders) | 32 (34) | 30 (44)
Oedema Peripheral (General disorders) | 18 (22) | 30 (38)
Pyrexia (General disorders) | 19 (21) | 22 (27)
Weight Decreased (Investigations) | 2 (3) | 10 (10)
Fall (Injury, poisoning and procedural complications) | 9 (11) | 11 (15)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 (1) | 52 (56)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2020-11-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT02990338/Prot_002.pdf
  • Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT02990338/SAP_003.pdf